CLINICAL TRIAL: NCT02361840
Title: Predictive Value of Troponin I for Acute Respiratory Distress Syndrome in Children With Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, KARLA ISIS AVILES MARTINEZ, MD Karla Isis Aviles Martinez, Hospital Civil de Guadalajara
Other Study IDs: HCFAA 003/12
Record Dates: First submitted 2014-12-31; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: ARDS
Keywords: Troponin I; Pediatric shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed cohort: TI>0.05ng/ml: We call Exposed group to increased TI > or = 0.05ng/ml We call Event to the onset of ARDS
- No Exposed cohort: TI<0.05ng/ml: We cal no Exposed group to increased TI (<0.05ng/ml) We call Event to the onset of ARDS

SUMMARY:
Shock is one of the five leading causes of income and mortality in emergencies. It generates a decrease in the availability of oxygen to the tissues, resulting in ischemia, pulmonary involvement and tissue reperfusion syndrome. This pathologies can trigger Syndrome of Acute Respiratory Distress (ARDS) and death.

Troponin I (TI) has been reported as early marker for ischemia and mortality other than coronary syndromes in critical patients.

Objective. Set the increase of TI as a predictor of ARDS in children with shock.

Null hypothesis. Increase serum in children with shock predicts the onset of ARDS.

Methodology. Prospective cohort type test diagnostic. Displays institutional. Sampling non-probability, consecutive inclusion. Calculation of the sample size: interval of confidence (IC) 95%, power - 80%; ratio non-exposed: exposed 2:1; n = 62.

Inclusion criteria: informed consent signed by the parent; children admitted to pediatric emergency (PEU) 1 month to 14 years with shock requiring mechanical ventilation.

Exclusion criteria: intake of toxic (TI value increment per will), ≥3 concentrated erythrocyte transfusion or plasma prior to entering PEU.

The investigators call exposure to the increase of TI≥0 05ng/ml and event to the development of ARDS. Determine TI value in plasma serum in the first 24 h, through Enzyme Immunoassay for the Quantitative Determination of Cardiac-Specific Troponin-I in Human Serum (cTnI ELISA), (reported as cardiac triage). Monitoring for 7 days.

Study was approved by Hospital Ethics Committee (Research record 003/12)

DETAILED DESCRIPTION:
INTRODUCTION The purpose of the present study is to establish a Troponin I (TI) in peripheral blood as a prognostic indicator in the emergence of the syndrome of acute respiratory difficulty (ARDS) in children with shock.

It should be noted that both shock and ARDS are life-threatening disease and one can trigger another (shock first then ARDS or ARDS then shock). Both involve abnormalities in blood flow (perfusion) tissues that leads to cellular stress, reduction of oxygen suplly (hypoxia), nutrients, consenquently generating an increase in tissue´s metabolic demands. This set of events is called ischemia.

The shock is a dynamic clinical syndrome of acute and complex circulatory dysfunction, caused by severe illness or trauma. To perpetuate itself generates multiple organ dysfunction and death. Regardless of its cause, it is conceptualized as a state of acute oxygen deficiency that prevents cell sustainability. The shock is one of the five leading causes of admission to emergency Pediatrics unit (EPU) of the Hospital Civil de Guadalajara "Fray Antonio Alcalde" (HCFAA).

Shock is the second cause of mortality in patients in the EPU. ARDS is an acute and diffuse, pulmonary inflammatory lesion characterized by increased pulmonary vascular permeability, weight and the decrease ventilation on the lung tissue. The specific clinical elements are hypoxemia and bilateral radiographic opacities associated with increases in the mixture of venous blood, physiological dead space and reduction of the pulmonary compliance. Diffuse alveolar damage is the morphological element that is in the acute phase (e.g. swelling, inflammation, hyaline membrane or bleeding). It has a mortality rate of 30-50% in the world.

TI is a protein that is determined in blood only under pathological conditions; mainly increases when there is myocardial ischemia. It was used in the first instance to diagnose acute coronary syndromes as ischemia, coronary angina pectoris and acute myocardial infarction.

It has been documented increase of TI in patients in critical condition without coronary disease, mainly in individuals with sepsis, septic shock, hypovolemic shock and children with respiratory failure by respiratory syncytial virus; in addition, has interpreted as a prognostic marker for mortality.

TI seems to anticipate the clinical signs of events persistent with hypoxia that may lead to ischemia. The elevation of serum levels of TI indicate myocardial damage, but they do not explain the underlying mechanism.

The addition of ARDS shock generates a troubling circumstance. However, not all children presentig shock develop ARDS; so it is necessary to predict ARDS or diagnose it in its earliest stage; This will impact on the implementation of strategies to avoid the severe form of the disease. With this foundation the investigators propose to use TI as a prognostic indicator of ARDS in children with shock.

To validate our hypothesis we conduct a study of dynamic and prospective cohort, type diagnostic test.

The exposed cohort is represented by children with shock that took TI increased during follow-up; of these patients was analyzed ARDS (event) who presented with TI high (exhibition) and those who develop ARDS with normal TI.

Determine a sample peripheral blood in the first 24 hours, taken from infants who presented shock without ARDS joining EPU sign consent of the parents who accepted the participation of children in the study.

The quantitative results of the sample are obtained by ELISA test sandwich with immunofluorescence, carried out in the Emergency Robotic laboratory of Robotics of the HCFAA. The investigators will monitor patients daily for 7 days; the data obtained will be documented on the blog for this purpose.

The investigators determine as exposure to the increase of TI with a serum value equal or greater than 0. 05ng/ml.

The investigators believe the development of ARDS event . The diagnosis of ARDS will be established in those children who met the criteria specified in the definition of Berlin for ARDS in 2012, within seven days after the onset shock.

The statistical analysis plan will consist in each case and as a whole, establish initial comparability of groups, will estimate the magnitude of the effect through partnership and finally, the investigators will make adjustments to the potential confounding factors.

The investigators will begin with descriptive statistics and will apply the Shapiro (for being a small sample) test to determine the normality of the distribution of the variables that define the type of statistical analysis to follow (parametric or free distribution).

Test Chi2 allows the comparison of proportions and risks for qualitative variables. Will use R Pearson or Spearman Rho tests to establish correlations between quantitative variables. Test Student's T or Mann-Whitney (according to the found data distribution) U will be used for the comparison of independent medium.

The investigators will consider significant value of p < 0.05.The estimate of the magnitude of the effect was carried out through determination of relative risk (RR) and absolute risk reduction (ARR).

The primary clinical research studies are represented by cross-sectional studies, cases and controls, cohort and clinical trials.

TI diagnostic test, we will calculate sensitivity, specificity, positive predictive value, negative predictive value, probability indexes and elaborate COR (Receiver Operating Characteristic) curve for optimum cutting of TI (quantitative variable expressed in ng/ml) to determine the approach of sensitivity and specificity.

QUESTION OF RESEARCH Does the increase in Troponin I serum in children with shock in Emergency Room can predict ARDS? General Objective. Establish increase TI value as a predictor of ARDS in children with shock.

Specific objectives. 1. To determine the incidence of children with shock that develops ARDS. 2. Establish correlation of TI with ARDS by Kirby oxygenation index. 3. To determine the sensitivity and specificity of TI in ARDS in children with shock. 4. Establish the serum prognostic value of TI for ARDS in children with shock The sample size Calculated sample size for study of prospective cohort with a confidence interval (CI) of 95%, 80% power. Exposed non-exposed 2:1 relation. Probability of occurring event in the cohort exposed 72% and 32% in the unexposed.

The investigators obtained 41 patients for unexposed cohort and 21 exposed are required to observe differences. Total number of 62 patients (n=62).

The sample size was calculated through the Epi Info version 7 of the Centers for Disease Control and Prevention (CDC), Atlanta.

Population Population was taken from the room of Emergency Pediatric Unit (EPU) of the Hospital Civil Fray Antonio Alcalde (HCFAA).

Inclusion criteria

1. Informed consent signed by the parent to participate in the study.
2. Children admitted to EPU of the HCFAA of 1 month old to 14 years old showing shock with less than 24 hour evolution.
3. Need for endotracheal intubation and mechanical ventilation. Exclusion criteria

1. Intake of toxic tricyclic antidepressants, cocaine and methamphetamines 2. Transfusion three or more concentrated erythrocyte / plasma before entering EPU.

3. Pregnant girls 4. Children with a previous diagnosis of uremic kidney injury. Criteria of elimination

1. Parents or legal guardians of patients requesting to leave the study.
2. Does not have gas analysis with lactate at the time of final categorization as shock.

Procedure The investigators included children with shock, categorized by instrument of Pediatric assessment consisting of General assessment, primary, secondary and tertiary assessment triangle.

The doctors who performed the final categorization of patients are pediatrician or pediatric residents certified under the American Academy of Pediatrics and the American Heart Association Pediatric Advanced Life Support.

Physicians were trained to one hour in pediatric evaluation and management of the instrument prior their participation. For this purpose, the instrument was the admission of Hospital Triage sheet. The possibilities of categorization initial pathophysiological according to the triangle of General evaluation are as follow:

1. Stable (three parts of the normal triangle)
2. Primary Disfunction of Central Nervous System or metabolic (abnormal appearance)
3. Shortness of breath (abnormal breathing)
4. Respiratory failure (abnormal breathing with abnormal color or appearance).
5. Shock (abnormal color)
6. Cardiorespiratory failure / imminent death (three parts of abnormal triangle) disease.

Immediately after categorization was a primary evaluation;was performed corresponding of a placement of monitor and measurement of vital signs, as well as evaluating and giving an A-B-C-D-E type treatment: air-permeable (A), control and management of the breath (B), circulation (C), identification of neurological Deficit (D) and (E) exhibition.

Within the laboratory studies requested in the tertiary evaluation, held gases in arterial blood lactate measurement.

If the children meet the inclusion criteria, they entered the cohort study. One mililiter of blood sample from the first 24 hours of the onset of shock was collected in a special tube containing anticoagulant and specially marked with a purple lid by its manufacturer.

The samples were taken to the emergency laboratory of the HCFAA within 10 minutes of obtaining them, they were processed using ELISA test sandwich by immunofluorescence using the reagent Enzyme Immunoassay for the Quantitative Determination of Cardiac-Specific Troponin-I in Human Serum (cTnI) ELISA.

The results were reported by the laboratory within 30 minutes after delivery, reported as cardiac Triage.

The result of TI is expressed as it is within range when the value is less than 0. 05ng/ml and high or out of range when the value is equal to or greater than 0. 05ng/ml. Once obtained the results, were added to the document in the protocol's log.

Stroke ECG and Echocardiogram was performed to all patients, conducted by an MD., Pediatrician Certified Cardiologist.

The patients were followed for 7 days from the entry to the cohort. The investigators have described as exposure for this cohort, TI ≥0. 05ng/ml increase and consider the development of ARDS, according to the definition of 2012 Berlin, even the latter constituted a measuring instrument.

There is no conflict of interest. Equipment and reagent for the determination of TI were obtained through public tender by the officer of Administrative Hospital Subdirector of HCFAA.

Dependent (outcome) variable: ARDS Independent (Predictor) variables: Troponin I

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the parent to participate in the study.
* Children admitted to EUP the HCFAA of 1 month old 14 years showing shock with less than 24 hour evolution.
* Need for endotracheal intubation and mechanical ventilation.

Exclusion Criteria:

* Intake of toxic tricyclic antidepressants, cocaine and methamphetamines that increase value of TI per se.
* Transfusion three or more concentrated erythrocyte / plasma before entering UP.
* Pregnant girls
* Children with a previous diagnosis of uremic kidney injury

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The sample size Calculated sample size for study of prospective cohort with a confidence interval (CI) of 95%, 80% power. Exposed non-exposed 2:1 relation. Probability of occurring event in the cohort exposed 72% and 32% in the unexposed.
  We calculated that 41 patients of unexposed cohort and 21 of the exposed are required to observed differences. Total number of 62 patients (n=62).
  The sample size was calculated through the Epi Info version 7 of the Centers for Disease Control and Prevention (CDC), Atlanta.
  Population Population was taken from the room of emergency Pediatrics of the Hospital Civil Fray Antonio Alcalde (HCFAA).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Determination of results of Primary study cohort | 2 years
  incidence of exposed , unexposed incidence , relative risk, attributable risk , absolute risk reduction

SECONDARY OUTCOMES:
Diagnostic Test | 2 months
  Sensibility, specificity, likelihoods ratio

CONTACTS AND LOCATIONS:
Overall Officials: KARLA ISIS AVILES MARTINEZ, MD, Principal Investigator — University of Guadalajara; MONICA CECILIA URIBE MERCADO, PhD., MD, Study Director — Universidad de Gudadalajara; IRAM ALBERTO VILLA MANZANO, PhD., MD, Study Director — University of Guadalajara
Locations (1):
- Karla Isis Aviles Martinez, Guadalajara, Jalisco, Mexico